CLINICAL TRIAL: NCT04674033
Title: The Sweet PEA Study: a Pilot Study of the Impact of Non-nutritive Sweetener Consumption During Pregnancy on Maternal and Infant Metabolic Health
Brief Title: The Sweet PEA Study: Effects of Diet During Pregnancy on Infant Growth and Development.
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Michael I. Goran, Principal Investigator, University of Southern California
Other Study IDs: CHLA-18-00455
Record Dates: First submitted 2020-12-08; First posted 2020-12-17 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Obesity
Keywords: Pregnancy; Nutrition; Obesity; Mother; Infant; Cognitive development; Growth
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Breast milk; Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Consumer: Participants who self-report regular consumption of non-nutritive sweeteners (>/=5 servings/week) based on a pre-screening dietary survey.
- Non-Consumer: Participants who self-report no consumption of non-nutritive sweeteners (0 servings/week) based on a pre-screening dietary survey.

SUMMARY:
The purpose of the Sweet PEA Study is to determine whether diet during pregnancy has an effect on infant's growth, body composition, and brain development.

DETAILED DESCRIPTION:
Rationale: Non-nutritive sweetener (NNS) consumption during pregnancy is prevalent, but effects on maternal and infant health are not well known. Intervention: None Objectives: To determine whether NNS consumption during pregnancy is associated with increased infant body fat, as well as differences in infant growth, brain structure/function, gut microbiota, and gestational diabetes. Study population: Women prior to 28 weeks' gestation, determined to have either low/no NNS consumption (control) or high NNS consumption (experimental), based on a pre-screening survey. Methodology: Identify two groups (low/high consumers) in early pregnancy, collect data during pregnancy remotely (telephone, internet, medical records) to determine diet and any link to pregnancy complications, have in-person visits with mothers/infants at 1, 6, and 12 months of age, collecting: body composition data (by EchoMRI), brain structure/connectivity (MRI), stool samples. Outcomes: Primary outcome is infant adiposity at 1, 6, and 12 months. Additional measures include infant growth, feeding behaviors, brain structure/ connectivity, gut microbiota, and maternal metabolic outcomes during routine gestational testing (fasting glucose, insulin, triglycerides, gestational diabetes diagnosis) Follow-up: This will operate as a small pilot study, and a larger study with more participants, a wider spectrum of NNS exposure, and longer follow up (into childhood and beyond) may follow. Statistics: Multivariate linear mixed effects examining maternal NNS intake and outcomes across time (repeated measures)

ELIGIBILITY:
Inclusion Criteria:

Mothers:

* Pregnant women prior to 28 weeks gestation
* Report the least NNS consumption of pre-screened participants (0 servings per week - representing the control group) and most NNS consumption of pre-screened participants (≥ 5 servings per week - representing the experimental group).
* 18-40 years of age
* Singleton pregnancy
* Be able/willing to understand the procedures of the study
* Be able to read English at a 5th grade level (materials also available in Spanish, if required)

Infants:

* Infant's mother must be enrolled in the study and provide infant assent to participate

Exclusion Criteria:

Mothers:

* Physician diagnosis of a major medical illness
* Pre-existing diabetes (type 1 or type 2), or GDM in a previous pregnancy
* Physical, mental, or cognitive issues preventing participation
* Medications that may affect body weight, body composition, insulin resistance, or lipid profiles
* Tobacco or drug use (any current use or quitting during pregnancy)
* Alcohol consumption during pregnancy (>1 drink per week)

Infants:

* Presumed or known congenital birth defects

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women (18 - 40 years) who do and do not report non-nutritive sweetener consumption, and their infants (<1-12 months) from Los Angeles, CA.
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Infant length at 1 Month | 1 month
  Infant length (cm) will be measured using an infant measure mat.
Infant length at 6 Months | 6 months
  Infant length (cm) will be measured using an infant measure mat.
Infant length at 12 Months | 12 months
  Infant length (cm) will be measured using an infant measure mat.
Infant weight at 1 Month | 1 month
  Infant weight (kg) will measured using a portable digital scale. For infants that need to be held, weight will be calculated as follows: (combined mother + infant weight) - (mother only weight).
Infant weight at 6 Months | 6 months
  Infant weight (kg) will measured using a portable digital scale. For infants that need to be held, weight will be calculated as follows: (combined mother + infant weight) - (mother only weight).
Infant weight at 12 Months | 12 months
  Infant weight (kg) will measured using a portable digital scale. For infants that need to be held, weight will be calculated as follows: (combined mother + infant weight) - (mother only weight).
Infant weight z-scores at 1 Month | 1 month
  Weight and length will be used to calculate weight-for-length (WLZ) and weight-for-age (WAZ) z-scores using the WHO Child Growth Standards, as recommended by the CDC for children <24 mos.
Infant weight z-scores at 6 Months | 6 months
  Weight and length will be used to calculate weight-for-length (WLZ) and weight-for-age (WAZ) z-scores using the WHO Child Growth Standards, as recommended by the CDC for children <24 mos.
Infant weight z-scores at 12 Months | 12 months
  Weight and length will be used to calculate weight-for-length (WLZ) and weight-for-age (WAZ) z-scores using the WHO Child Growth Standards, as recommended by the CDC for children <24 mos.
Infant body fat measured using an EchoMRI body composition analyzer at 1 month | 1 month
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant body fat in grams.
Infant body fat measured using an EchoMRI body composition analyzer at 6 months | 6 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant body fat in grams.
Infant body fat measured using an EchoMRI body composition analyzer at 12 months | 12 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant body fat in grams.
Infant lean mass measured using an EchoMRI body composition analyzer at 1 month | 1 month
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant lean mass in grams.
Infant lean mass measured using an EchoMRI body composition analyzer at 6 months | 6 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant lean mass in grams.
Infant lean mass measured using an EchoMRI body composition analyzer at 12 months | 12 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant lean mass in grams.
Infant total body water measured using an EchoMRI body composition analyzer at 1 month | 1 month
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant total body water in grams.
Infant total body water measured using an EchoMRI body composition analyzer at 6 months | 6 month
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant total body water in grams.
Infant total body water measured using an EchoMRI body composition analyzer at 12 months | 12 month
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant total body water in grams.
Infant free body water measured using an EchoMRI body composition analyzer at 1 month | 1 month
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant free body water in grams.
Infant free body water measured using an EchoMRI body composition analyzer at 6 months | 6 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant free body water in grams.
Infant free body water measured using an EchoMRI body composition analyzer at 12 months | 12 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant free body water in grams.

SECONDARY OUTCOMES:
Maternal height at 1 month | 1 month
  Height (cm) will be measured using a stadiometer.
Maternal height at 6 months | 6 months
  Height (cm) will be measured using a stadiometer.
Maternal height at 12 months | 12 months
  Height (cm) will be measured using a stadiometer.
Maternal weight at 1 month | 1 month
  Weight (kg) will be measured using a portable digital scale.
Maternal weight at 6 months | 6 months
  Weight (kg) will be measured using a portable digital scale.
Maternal weight at 12 months | 12 months
  Weight (kg) will be measured using a portable digital scale.
Maternal BMI at 1 Month | 1 month
  Body Mass Index (BMI) will be calculated based on the equation (weight in kg)/(height in m)^2.
Maternal BMI at 6 Months | 6 months
  Body Mass Index (BMI) will be calculated based on the equation (weight in kg)/(height in m)^2.
Maternal BMI at 12 Months | 12 months
  Body Mass Index (BMI) will be calculated based on the equation (weight in kg)/(height in m)^2.
Maternal blood glucose at Pregnancy visit 2 | ~35 weeks' gestation
  Mothers will self-report their most recent blood glucose levels.
Maternal pregravid BMI | 24-28 weeks' gestation
  Maternal BMI prior to pregnancy will be derived from pregravid BMI (recall during pregnancy) using the equation (weight in kg)/(height in m)^2.
Maternal blood pressure at 1 month | 1 month
  Sitting blood pressure will be measured on the right arm after the subject has rested quietly for 5 minutes using a digital blood pressure monitor (Omron 3-series).
Maternal blood pressure at 6 months | 6 months
  Sitting blood pressure will be measured on the right arm after the subject has rested quietly for 5 minutes using a digital blood pressure monitor (Omron 3-series).
Maternal blood pressure at 12 months | 12 months
  Sitting blood pressure will be measured on the right arm after the subject has rested quietly for 5 minutes using a digital blood pressure monitor (Omron 3-series).
Maternal resting heart rate at 1 month | 1 month
  Sitting heart rate will be measured on the right arm after the subject has rested quietly for 5 minutes using a digital blood pressure monitor (Omron 3-series).
Maternal resting heart rate at 6 months | 6 months
  Sitting heart rate will be measured on the right arm after the subject has rested quietly for 5 minutes using a digital blood pressure monitor (Omron 3-series).
Maternal resting heart rate at 12 months | 12 months
  Sitting heart rate will be measured on the right arm after the subject has rested quietly for 5 minutes using a digital blood pressure monitor (Omron 3-series).
Maternal diet at Pregnancy visit 1 | 24-28 weeks' gestation
  24-hour diet recalls will be conducted for one week day and one weekend day. Dietary intake will be collected and analyzed using the most current version of the Nutrition Data System for Research software (NDSR).
Maternal diet at Pregnancy visit 2 | ~35 weeks' gestation
  24-hour diet recalls will be conducted for one week day and one weekend day. Dietary intake will be collected and analyzed using the most current version of the Nutrition Data System for Research software (NDSR).
Maternal diet at 1 month | 1 month
  24-hour diet recalls will be conducted for one week day and one weekend day. Dietary intake will be collected and analyzed using the most current version of the Nutrition Data System for Research software (NDSR).
Maternal diet at 6 months | 6 months
  24-hour diet recalls will be conducted for one week day and one weekend day. Dietary intake will be collected and analyzed using the most current version of the Nutrition Data System for Research software (NDSR).
Maternal diet at 12 months | 12 months
  24-hour diet recalls will be conducted for one week day and one weekend day. Dietary intake will be collected and analyzed using the most current version of the Nutrition Data System for Research software (NDSR).
Infant diet at 1 month | 1 month
  24-hour diet recalls will be conducted for one week day and one weekend day. Mothers will be interviewed to report on their infant's food intake. Dietary intake will be collected and analyzed using the most current version of the Nutrition Data System for Research software (NDSR).
Infant diet at 6 months | 6 months
  24-hour diet recalls will be conducted for one week day and one weekend day. Mothers will be interviewed to report on their infant's food intake. Dietary intake will be collected and analyzed using the most current version of the Nutrition Data System for Research software (NDSR).
Infant diet at 12 months | 12 months
  24-hour diet recalls will be conducted for one week day and one weekend day. Mothers will be interviewed to report on their infant's food intake. Dietary intake will be collected and analyzed using the most current version of the Nutrition Data System for Research software (NDSR).
Infant feeding score assessed by Infant Feeding Questionnaire at 1 month | 1 month
  Infant feeding score will be assessed using the Baughcum Infant Feeding Questionnaire. Questions are scored using the following scale: 1-5; never, rarely, sometimes, often, always. Average scores will be used to determine the following constructs: concern about the child undereating or becoming underweight; concern about infant's hunger; awareness of infant's cues; concern about the infant becoming overweight or overeating; feeding the infant on schedule; using food to calm the infant; social interaction during feeding.
Infant feeding score assessed by Infant Feeding Questionnaire at 6 months | 6 months
  Infant feeding score will be assessed using the Baughcum Infant Feeding Questionnaire. Questions are scored using the following scale: 1-5; never, rarely, sometimes, often, always. Average scores will be used to determine the following constructs: concern about the child undereating or becoming underweight; concern about infant's hunger; awareness of infant's cues; concern about the infant becoming overweight or overeating; feeding the infant on schedule; using food to calm the infant; social interaction during feeding.
Infant feeding score assessed by Infant Feeding Questionnaire at 12 months | 12 months
  Infant feeding score will be assessed using the Baughcum Infant Feeding Questionnaire. Questions are scored using the following scale: 1-5; never, rarely, sometimes, often, always. Average scores will be used to determine the following constructs: concern about the child undereating or becoming underweight; concern about infant's hunger; awareness of infant's cues; concern about the infant becoming overweight or overeating; feeding the infant on schedule; using food to calm the infant; social interaction during feeding.
Infant feeding style score assessed by Infant Feeding Style Questionnaire at 1 month | 1 month
  Infant feeding style score will be assessed using the Thompson Infant Feeding Style Questionnaire. Questions are scored using the following scale: 1-5; disagree, slightly disagree, neutral, slightly agree, agree. Average scores will be used to determine the following constructs: laissez-faire; pressuring; restrictive; responsive; and indulgent.
Infant feeding style score assessed by Infant Feeding Style Questionnaire at 6 months | 6 months
  Infant feeding style score will be assessed using the Thompson Infant Feeding Style Questionnaire. Questions are scored using the following scale: 1-5; disagree, slightly disagree, neutral, slightly agree, agree. Average scores will be used to determine the following constructs: laissez-faire; pressuring; restrictive; responsive; and indulgent.
Infant feeding style score assessed by Infant Feeding Style Questionnaire at 12 months | 12 months
  Infant feeding style score will be assessed using the Thompson Infant Feeding Style Questionnaire. Questions are scored using the following scale: 1-5; disagree, slightly disagree, neutral, slightly agree, agree. Average scores will be used to determine the following constructs: laissez-faire; pressuring; restrictive; responsive; and indulgent.
Infant behavior score assessed by Infant Behavior Questionnaire at 1 month | 1 month
  Infant behavior score will be assessed using the Rothbart Infant Behavior Questionnaire. Questions are scored using the following scale: 1-7; never, very rarely, less than half the time, about half the time, more than half the time, almost always, always. Composite scores will be used to determine the following constructs: surgency/extroversion; negative affectivity; and orienting/regulation.
Infant behavior score assessed by Infant Behavior Questionnaire at 6 months | 6 months
  Infant behavior score will be assessed using the Rothbart Infant Behavior Questionnaire. Questions are scored using the following scale: 1-7; never, very rarely, less than half the time, about half the time, more than half the time, almost always, always. Composite scores will be used to determine the following constructs: surgency/extroversion; negative affectivity; and orienting/regulation.
Infant behavior score assessed by Infant Behavior Questionnaire at 12 months | 12 months
  Infant behavior score will be assessed using the Rothbart Infant Behavior Questionnaire. Questions are scored using the following scale: 1-7; never, very rarely, less than half the time, about half the time, more than half the time, almost always, always. Composite scores will be used to determine the following constructs: surgency/extroversion; negative affectivity; and orienting/regulation.
Infant eating behavior score assessed by Baby Eating Behavior Questionnaire at 1 month | 1 month
  Infant eating behavior score will be assessed using the Llewellyn Baby Eating Behavior Questionnaire. Questions are scored using the following scale: 1-5; never, rarely, sometimes, often, always. Average scores will be used to determine the following constructs: food responsiveness; satiety responsiveness; slowness in eating; enjoyment of food; and general appetite.
Infant eating behavior score assessed by Baby Eating Behavior Questionnaire at 6 months | 6 months
  Infant eating behavior score will be assessed using the Llewellyn Baby Eating Behavior Questionnaire. Questions are scored using the following scale: 1-5; never, rarely, sometimes, often, always. Average scores will be used to determine the following constructs: food responsiveness; satiety responsiveness; slowness in eating; enjoyment of food; and general appetite.
Infant eating behavior score assessed by Baby Eating Behavior Questionnaire at 12 months | 12 months
  Infant eating behavior score will be assessed using the Llewellyn Baby Eating Behavior Questionnaire. Questions are scored using the following scale: 1-5; never, rarely, sometimes, often, always. Average scores will be used to determine the following constructs: food responsiveness; satiety responsiveness; slowness in eating; enjoyment of food; and general appetite.
Breast milk composition at 1 month | 1 month
  Breast milk will be collected from mothers at least 11⁄2 hours since the last feeding and while the mother has fasted at least 1 hour. Samples will be analyzed for glucose, fructose, galactose, lactose and sucrose by mass spectrometry. Samples will be available for analysis of insulin, leptin, and energy content.
Breast milk composition at 6 months | 6 months
  Breast milk will be collected from mothers at least 11⁄2 hours since the last feeding and while the mother has fasted at least 1 hour. Samples will be analyzed for glucose, fructose, galactose, lactose and sucrose by mass spectrometry. Samples will be available for analysis of insulin, leptin, and energy content.
Breast milk composition at 12 months | 12 months
  Breast milk will be collected from mothers at least 11⁄2 hours since the last feeding and while the mother has fasted at least 1 hour. Samples will be analyzed for glucose, fructose, galactose, lactose and sucrose by mass spectrometry. Samples will be available for analysis of insulin, leptin, and energy content.
Infant Magnetic Resonance Imaging (MRI) brain scan at 1 month | 1 month
  Infant brain will be scanned using Magnetic Resonance Imaging (MRI) to measure structure and function.
Infant Magnetic Resonance Imaging (MRI) brain scan at 6 months | 6 months
  Infant brain will be scanned using Magnetic Resonance Imaging (MRI) to measure structure and function.
Infant gut microbiome at 1 Month | 1 month
  Stool samples will be collected in OmniGUT gene kits and aliquoted to be stored at -80oC. Gut microbes will be analyzed using 16S sequencing.
Infant gut microbiome at 6 Months | 6 months
  Stool samples will be collected in OmniGUT gene kits and aliquoted to be stored at -80oC. Gut microbes will be analyzed using 16S sequencing.
Infant gut microbiome at 12 Months | 12 months
  Stool samples will be collected in OmniGUT gene kits and aliquoted to be stored at -80oC. Gut microbes will be analyzed using 16S sequencing.
Maternal gut microbiome at 1 month | 1 month
  Stool samples will be collected in OmniGUT gene kits and aliquoted to be stored at -80oC. Gut microbes will be analyzed using 16S sequencing.
Maternal gut microbiome at 6 months | 6 months
  Stool samples will be collected in OmniGUT gene kits and aliquoted to be stored at -80oC. Gut microbes will be analyzed using 16S sequencing.
Maternal gut microbiome at 12 months | 12 months
  Stool samples will be collected in OmniGUT gene kits and aliquoted to be stored at -80oC. Gut microbes will be analyzed using 16S sequencing.
Infant Diet and Behavior Questionnaire at 1 month | 1 month
  Participants will report when they stopped breastfeeding/introduced formula or solid foods.
Infant Diet and Behavior Questionnaire at 6 months | 6 months
  Participants will report when they stopped breastfeeding/introduced formula or solid foods.
Infant Diet and Behavior Questionnaire at 12 months | 12 months
  Participants will report when they stopped breastfeeding/introduced formula or solid foods.
CDC Infant Feeding Practices Survey II at 1 month | 1 month
  Participants will answer questions about their and their infant's diet.
CDC Infant Feeding Practices Survey II at 6 months | 6 months
  Participants will answer questions about their and their infant's diet.
CDC Infant Feeding Practices Survey II at 12 months | 12 months
  Participants will answer questions about their and their infant's diet.
Maternal Beverage Recall at Pregnancy visit 1 | 24-28 weeks' gestation
  Participants will report the beverages they have consumed over the past week. This data will be used to assess nutritional intake based on beverages.
Maternal Beverage Recall at Pregnancy visit 2 | ~35 weeks' gestation
  Participants will report the beverages they have consumed over the past week. This data will be used to assess nutritional intake based on beverages.
Maternal Beverage Recall at 1 month | 1 month
  Participants will report the beverages they have consumed over the past week. This data will be used to assess nutritional intake based on beverages.
Maternal Beverage Recall at 6 months | 6 months
  Participants will report the beverages they have consumed over the past week. This data will be used to assess nutritional intake based on beverages.
Maternal Beverage Recall at 12 months | 12 months
  Participants will report the beverages they have consumed over the past week. This data will be used to assess nutritional intake based on beverages.
Infant Beverage Recall at 1 month | 1 month
  Mother's will report the beverages their infant has consumed over the past week. This data will be used to assess nutritional intake based on beverages.
Infant Beverage Recall at 6 months | 6 months
  Mother's will report the beverages their infant has consumed over the past week. This data will be used to assess nutritional intake based on beverages.
Infant Beverage Recall at 12 months | 12 months
  Mother's will report the beverages their infant has consumed over the past week. This data will be used to assess nutritional intake based on beverages.
Perinatal Anxiety Screening Scale (PASS) at Pregnancy visit 1 | 24-28 weeks' gestation
  Participants will answer questions regarding their stress levels during and after pregnancy. Minimum = 0; maximum = 93. Higher scores represent worse outcomes.
Perinatal Anxiety Screening Scale (PASS) at Pregnancy visit 2 | ~35 weeks' gestation
  Participants will answer questions regarding their stress levels during and after pregnancy. Minimum = 0; maximum = 93. Higher scores represent worse outcomes.
Perinatal Anxiety Screening Scale (PASS) at 1 month | 1 month
  Participants will answer questions regarding their stress levels during and after pregnancy. Minimum = 0; maximum = 93. Higher scores represent worse outcomes.
Perinatal Anxiety Screening Scale (PASS) at 6 months | 6 months
  Participants will answer questions regarding their stress levels during and after pregnancy. Minimum = 0; maximum = 93. Higher scores represent worse outcomes.
Perinatal Anxiety Screening Scale (PASS) at 12 months | 12 months
  Participants will answer questions regarding their stress levels during and after pregnancy. Minimum = 0; maximum = 93. Higher scores represent worse outcomes.
Edinburgh Postnatal Depression Scale (EPDS) at Pregnancy visit 1 | 24-28 weeks' gestation
  Participants will answer questions regarding their feelings and mood. Minimum = 0, maximum = 30. Higher scores represent worse outcomes.
Edinburgh Postnatal Depression Scale (EPDS) at Pregnancy visit 2 | ~35 weeks' gestation
  Participants will answer questions regarding their feelings and mood. Minimum = 0, maximum = 30. Higher scores represent worse outcomes.
Edinburgh Postnatal Depression Scale (EPDS) at 1 month | 1 month
  Participants will answer questions regarding their feelings and mood. Minimum = 0, maximum = 30. Higher scores represent worse outcomes.
Edinburgh Postnatal Depression Scale (EPDS) at 6 months | 6 months
  Participants will answer questions regarding their feelings and mood. Minimum = 0, maximum = 30. Higher scores represent worse outcomes.
Edinburgh Postnatal Depression Scale (EPDS) at 12 months | 12 months
  Participants will answer questions regarding their feelings and mood. Minimum = 0, maximum = 30. Higher scores represent worse outcomes.
Pregnancy Physical Activity Questionnaire at Pregnancy visit 1 | 24-28 weeks' gestation
  Participants will answer questions about their physical activity levels over the past week. Minimum: 0 (none), maximum: 5 (3 or more hours per day). Higher scores represent better outcomes.
Pregnancy Physical Activity Questionnaire at Pregnancy visit 2 | ~35 weeks' gestation
  Participants will answer questions about their physical activity levels over the past week. Minimum: 0 (none), maximum: 5 (3 or more hours per day). Higher scores represent better outcomes.
Pregnancy Physical Activity Questionnaire at 1 month | 1 month
  Participants will answer questions about their physical activity levels over the past week. Minimum: 0 (none), maximum: 5 (3 or more hours per day). Higher scores represent better outcomes.
Pregnancy Physical Activity Questionnaire at 6 months | 6 months
  Participants will answer questions about their physical activity levels over the past week. Minimum: 0 (none), maximum: 5 (3 or more hours per day). Higher scores represent better outcomes.
Pregnancy Physical Activity Questionnaire at 12 months | 12 months
  Participants will answer questions about their physical activity levels over the past week. Minimum: 0 (none), maximum: 5 (3 or more hours per day). Higher scores represent better outcomes.
Pittsburgh Sleep Quality Index (PSQI) at Pregnancy visit 1 | 24-28 weeks' gestation
  Participants will answer questions about their sleeping habits over the past week.
Pittsburgh Sleep Quality Index (PSQI) at Pregnancy visit 2 | ~35 weeks' gestation
  Participants will answer questions about their sleeping habits over the past week.
Pittsburgh Sleep Quality Index (PSQI) at 1 month | 1 month
  Participants will answer questions about their sleeping habits over the past week.
Pittsburgh Sleep Quality Index (PSQI) at 6 months | 6 months
  Participants will answer questions about their sleeping habits over the past week.
Pittsburgh Sleep Quality Index (PSQI) at 12 months | 12 months
  Participants will answer questions about their sleeping habits over the past week.

CONTACTS AND LOCATIONS:
Overall Officials: Michael I Goran, Principal Investigator — University of Southern California; Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States